CLINICAL TRIAL: NCT07326332
Title: Effect of Dexmedetomidine Sedation on Tear Film in Patients Undergoing Angioplasty Under Local Anesthesia
Brief Title: Effect of Dexmedetomidine on Tear Production in Angioplasty Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Samar Rafik Mohamed Amin, Assistant professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RC.18.10.2025
Record Dates: First submitted 2025-12-16; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Tear Film Alteration
MeSH Terms: interventions — Dexmedetomidine; Midazolam; Fentanyl; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine Sedation (Experimental): Participants in this arm will be sedated with intravenous dexmedetomidine during angioplasty performed under local anesthesia. Dexmedetomidine will be administered as a loading dose (if clinically appropriate) followed by a continuous infusion titrated to achieve moderate sedation (RASS -2 to 0). Rescue sedation with small propofol boluses may be used if needed and will be recorded.
  Interventions: Drug: Dexmedetomidine
- Standard Sedation (Active Comparator): Participants in this arm will receive standard sedation according to routine clinical practice during angioplasty under local anesthesia. Sedation may include intermittent intravenous boluses of midazolam with or without opioid analgesics (e.g., fentanyl) and/or small propofol boluses, titrated to achieve moderate sedation (RASS -2 to 0).
  Interventions: Drug: Sedation with Midazolam, Fentanyl, and Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine will be administered intravenously for procedural sedation during angioplasty under local anesthesia. A loading dose of 0.4-0.6 µg/kg may be given over 10 minutes at the discretion of the anesthesiologist, followed by a continuous infusion of 0.2-0.7 µg/kg/hour titrated to achieve moderate sedation (RASS -2 to 0). Rescue sedation with small propofol boluses may be used if required and will be documented.
  Arms: Dexmedetomidine Sedation
Drug: Sedation with Midazolam, Fentanyl, and Propofol — Standard sedation will be provided according to routine clinical practice during angioplasty under local anesthesia. Sedation may include intermittent intravenous boluses of midazolam, with or without opioid analgesics (e.g., fentanyl), and/or small propofol boluses, titrated to achieve moderate sedation (RASS -2 to 0). All administered drugs and cumulative doses will be recorded.
  Arms: Standard Sedation

SUMMARY:
During medical procedures performed under local anesthesia with sedation, such as angioplasty, the eyes may become dry because normal blinking and tear production can be reduced. Dexmedetomidine is a commonly used sedative that provides comfort and pain relief while allowing patients to breathe on their own. However, there is limited information about how dexmedetomidine affects tear production and eye comfort after procedures.

This study aims to evaluate whether sedation with dexmedetomidine affects tear production compared with standard sedative medications used during angioplasty. Adult patients undergoing angioplasty under local anesthesia will be randomly assigned to receive either dexmedetomidine sedation or standard sedation. Tear production will be measured using the Schirmer test before the procedure, shortly after the procedure, and 12 hours later. Patients will also be asked about eye dryness or discomfort, and any eye-related or sedation-related side effects will be recorded.

The results of this study may help improve eye safety and comfort in patients receiving sedation during angioplasty and guide the selection of sedative medications in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective angioplasty (coronary PCI or peripheral angioplasty) under local anesthesia with planned procedural sedation.
* Able to give informed consent and complete ocular symptom assessments.
* Baseline Schirmer I ≥1 mm (to exclude complete anatomic lacrimal failure; you may alter this cutoff).

Exclusion Criteria:

* Pre-existing moderate/severe dry eye disease or Sjögren's syndrome (history or OSDI >33).
* Ocular surgery within prior 3 months or active ocular infection.
* Contact lens use within 24 hours before baseline.
* Chronic systemic medications known to substantially alter lacrimation (recent anticholinergics, high-dose tricyclics) unless stable and documented.
* Known allergy to dexmedetomidine, midazolam, fentanyl, or propofol.
* Significant bradycardia (HR <50) or high-degree AV block without pacemaker.
* Pregnancy or breastfeeding.
* Any condition making study participation or follow-up impossible.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Change in Tear Production Measured by Schirmer I Test | Baseline (30 minutes pre-procedure) to 30 minutes post-procedure
  Change in tear production measured by the Schirmer I test (without topical anesthesia), calculated as the difference in millimeters (mm) between baseline (pre-procedure, awake) and immediate post-procedure measurement once the patient is responsive (Aldrete score ≥9). Measurements will be performed in a standardized manner by a trained, blinded assessor.

SECONDARY OUTCOMES:
Immediate Post-Procedure Tear Production (Schirmer I Test) | 30-60 minutes after completion of the procedure
  Tear production measured using the Schirmer I test (mm) immediately after the procedure, once the patient is responsive (Aldrete score ≥9), and compared between study groups.
Patient-Reported Dry Eye Symptoms | Baseline (pre-procedure), immediate post-procedure, and 12 hours post-procedure
  Dry eye symptoms assessed using a visual analog scale (VAS) ranging from 0 to 10, where 0 = no dry eye symptoms and 10 = worst imaginable dry eye symptoms.
Incidence of Ocular Adverse Events | From start of procedure to 12 hours post-procedure
  Occurrence of ocular adverse events, including corneal abrasion, corneal epithelial defects, conjunctival hyperemia, blurred vision, or severe dry eye requiring ophthalmologic consultation.
Total Dexmedetomidine Dose | During the procedure
  Total cumulative dose of dexmedetomidine administered during the procedure, expressed in micrograms (µg).

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University Hospital, Banhā, Qalyubia Governorate, Egypt